CLINICAL TRIAL: NCT00857194
Title: Risk Factors for Coronary Heart Disease in Spinal Cord Injury: Conventional and Emerging
Brief Title: Cardiovascular Disease Study
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: B4162C-5
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Spinal Cord Injury
Keywords: Coronary Heart Disease; spinal cord injury; risk factor; postprandial lipemia
MeSH Terms: conditions — Spinal Cord Injuries; Coronary Disease | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 2: Chronic, stable spinal cord injury
  Interventions: Procedure: 2 hour Oral Glucose Tolerance Test; Procedure: Fat Meal Test

INTERVENTIONS:
Procedure: 2 hour Oral Glucose Tolerance Test — Fasting baseline blood samples will be drawn for analysis of insulin and glucose. A 75-gram glucose solution will be administered and subjects remain sedentary for 2 hours. After 2 hours, blood is drawn to analyze post-load insulin and glucose levels.
  Other Names: 2-hr OGTT
Procedure: Fat Meal Test — A fasting blood draw is performed for analysis of lipids, insulin, and glucose. Subjects ingest a high fat meal (milkshake made from heavy whipping cream and premium ice cream) within 15 minutes. Postprandial blood draws at 2, 4, and 6 hours are made for analysis of lipids, insulin, and glucose.

SUMMARY:
Coronary heart disease (CHD) is a leading cause of death in the spinal cord injured (SCI) population, occurring at younger ages than in the able-bodied population. Conventional risk factors for CHD include high concentrations of low-density lipoprotein (LDL), low concentrations of high-density lipoprotein (HDL), diabetes mellitus (DM), smoking history, and family history. Other factors that may influence progression of CHD include C-reactive protein (an inflammatory marker), and fibrinogen (a pro-coagulant marker). Individuals with SCI with longer duration and greater completeness of injury are more likely to have significantly worse carbohydrate tolerance compared to other neurological deficit subgroups. Muscle atrophy after SCI is associated with increased insulin resistance. Prolonged inactivity has been shown to be associated with hyperinsulinemia and impaired glucose tolerance. Body composition changes after SCI to indicate significantly more total body fat mass and percent fat and less lean mass compared to able-bodied individuals. Carotid intima-media thickness is correlated with atherosclerosis progression and abdominal adiposity. Individuals with abdominal adiposity are at a higher risk for CHD, DM, hypertension, insulin resistance, and dyslipidemia. Abdominal adiposity and insulin resistance are contributors to postprandial lipemia, which may be a more sensitive indicator of CHD risk and progression.

The purpose of this study is to determine the prevalence of conventional risk factors by assessing the 10-year risk for CHD, and identify emerging risk factors for CHD in the spinal cord injured population. Subjects will have the option to participate in a high fat meal test to determine postprandial lipemic responses. Knowledge of this information may be able to detect and prevent future cardiovascular events related to CHD.

ELIGIBILITY:
Inclusion Criteria:

* Male 45-75 years old with at least 5 years of SCI
* Female 45-50 years old with at least 10 years of SCI
* Female 50-75 years old with at least 5 years of SCI

Exclusion Criteria:

* Acute medical illness
* Pregnant females
* Chronic debilitating disease (i.e., heart disease, pulmonary disease, etc.)
* Atrial fibrillation
* History of percutaneous coronary angiography with stent placement

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from hospital clinics, through advertisements, and referral from primary care physicians.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
coronary heart disease risk factors | 1 time, at time of testing
  Risk factors associated with coronary heart disease as follows:
  * Fasting Lipid Panel
  * Oral Glucose Tolerance Test
  * Blood Pressure
  * Body Anthropometrics
  * Family History

SECONDARY OUTCOMES:
postprandial lipemic response to a high-fat meal | baseline, 2, 4, and 6 hrs post high fat meal
  Blood draws following ingestion of high fat meal at 2, 4, and 6 hours to determine lipids.

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Undecided